CLINICAL TRIAL: NCT03990675
Title: Evaluation and Comparison of the Growth Rate of Pancreatic Cancer Patient-derived Organoids Generated From Matched Fine Needle Aspirations (FNA) and Fine Needle Biopsies (FNB)
Brief Title: Evaluation and Comparison of the Growth Rate of Pancreatic Cancer Patient-derived Organoids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pancreatic cancer organoids
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Pancreas Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FNA, FNB (Experimental)
  Interventions: Procedure: FNA, FNB

INTERVENTIONS:
Procedure: FNA, FNB — Endoscopic ultrasound guided fine needle aspiration, Endoscopic ultrasound guided fine needle biopsy

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) is one of the most aggressive forms of cancer. Despite advances in the understanding of the mechanisms underlying PDAC pathogenesis, the impact on patient benefit is lagging. As a result, new model systems are being developed and used to fill this gap with the hope of translation into improved diagnostics and therapeutics.

Organoids represent a powerful tool for research with the capacity to be applied to many key aspects of pancreatic tissue pathology.

3D organoids can be generated from endoscopic fine-needle aspiration or fine needle biopsy samples. In this study, we will evaluate and compare the growth rate of pancreatic cancer patient-derived organoids generated from matched fine needle Aspirations (FNA) and fine needle biopsies (FNB).

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for EUS-guided FNA or FNB of a suspected pancreatic malignancy

Exclusion Criteria:

* < 18 years
* patients unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Growth rate | 4 days
  Organoid growth will be determined using bi-weekly measurements by phase-contrast microscopy calculating the total organoid area as well as individual organoid size. In addition, growth rates will be determined using the cell glow assay (Promega) over a time-course of 4 days. Furthermore, the mean passaging time will be calculated after 5 passages.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Medical Department, Klinikum rechts der Isar, Munich, Germany